CLINICAL TRIAL: NCT01126788
Title: Comparative Physiologic Technology Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Glenn LaMuraglia, MD, Massachusetts General Hospital
Other Study IDs: 2009P002554
Record Dates: First submitted 2010-05-18; First posted 2010-05-20 (Estimated); Last update posted 2010-11-24 (Estimated); Status verified 2010-11

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PADnet + testing
- Parks Flo-lab Test

SUMMARY:
This study is designed to test two hypotheses:

1. The PADnet+ testing system produces clinically equivalent results as the Parks Flo-Lab testing system in a group of patients referred for evaluation of PAD of the limbs when performed by a Registered Vascular Technologist (RVT).
2. The PADnet+ testing system produces clinically equivalent results when the testing is repeated on the above patients and performed by staff specifically trained on the use of the PADnet+ system but are not vascular technologists nor hold the RVT certification.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred to the MGH Vascular Labs for diagnostic testing for PAD

Exclusion Criteria:

* None

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred to the MGH Vascular Labs for diagnostic testing for PAD
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn LaMuraglia, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachsetts General Hospital, Boston, Massachusetts, United States